CLINICAL TRIAL: NCT07255573
Title: Diagnostic Accuracy of The Water Immersion Wrinkle Test for the Diagnosis of Small Fiber Neuropathy
Brief Title: Diagnostic Accuracy of The Water Immersion Wrinkle Test for Small Fiber Neuropathy
Acronym: WIWT-SFN
Status: Completed | Type: Observational
Sponsor: HOSPITAL BRITANICO DE BUENOS AIRES (Other)
Responsible Party: Principal Investigator, Lucas Piedrafita Vico, Principal Investigator, HOSPITAL BRITANICO DE BUENOS AIRES
Other Study IDs: 14202
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Small-Fiber Neuropathy; Dysautonomia
Keywords: small-fiber neuropathy; dysautonomia; water-immersion wrinkle test; QST; SSR
MeSH Terms: conditions — Small Fiber Neuropathy; Autonomic Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SFN Group: Adults evaluated in a tertiary neuromuscular clinic who, after baseline assessment, are classified as having small-fiber neuropathy (SFN) by the prespecified composite reference standard. The reference integrates (1) neuromuscular specialist clinical judgment (history and focused examination) and (2) abnormality on ≥1 validated scale (UENS or mTCNS) using published scoring rules. Group assignment is independent of WIWT, QST, or SSR results; these tests may be performed as index/comparator procedures but do not define cohort membership.
- Control Group: Adults evaluated in a tertiary neuromuscular clinic who, after baseline assessment, are classified as No Small-Fiber Neuropathy (No SFN) by the prespecified composite reference. This cohort includes healthy adult volunteers with no neuropathic symptoms or signs, a normal neurological examination, and normal UENS and mTCNS scores per published rules. Group assignment is independent of WIWT, QST, or SSR results; these tests may be performed as index/comparator procedures but do not define cohort membership.

SUMMARY:
Small-fiber neuropathy (SFN) affects A-delta and C fibers and commonly presents with sensory symptoms and dysautonomia. Confirmation often relies on specialized tests such as quantitative sensory testing (QST) and sympathetic skin response (SSR). This prospective, single-center observational diagnostic-accuracy study will estimate the performance of the Water-Immersion Wrinkle Test (WIWT) for detecting SFN in adults evaluated by a neuromuscular service. The composite reference standard is specialist clinical assessment plus abnormality on ≥1 validated scale (Utah Early Neuropathy Scale [UENS] or modified Toronto Clinical Neuropathy Score [mTCNS]). The index procedure (WIWT) is standardized as follows: both hands immersed to at least the distal interphalangeal crease for 15 minutes; immersion begins at 43-44 °C with expected passive cooling of ~2 °C every 5 minutes; temperature measured at 0, 5, 10 and 15 minutes; no water is added or replaced during immersion. After gentle drying, standardized photographs are obtained and wrinkling grades (0-4) are recorded for digits 2-5; the bilateral summed score is classified abnormal <24 and normal ≥24. Examiners for WIWT, QST, and SSR are mutually blinded. The primary outcome is WIWT sensitivity and specificity versus the composite reference at baseline. Secondary outcomes include ROC area under the curve (AUC), positive/negative predictive values, and inter- and intra-rater reliability (intraclass correlation coefficients). Recruitment is ongoing; anticipated primary completion: November 2025.

DETAILED DESCRIPTION:
This is a prospective, single-center, observational diagnostic-accuracy study designed to estimate the performance of the Water-Immersion Wrinkle Test (WIWT) for identifying small-fiber neuropathy (SFN) in adults evaluated by a neuromuscular department. The composite reference standard is a specialist clinical assessment consistent with SFN together with abnormality on at least one validated clinical scale (Utah Early Neuropathy Scale [UENS] or modified Toronto Clinical Neuropathy Score [mTCNS]). Quantitative Sensory Testing (QST) and Sympathetic Skin Response (SSR) are obtained as comparator tests but do not form part of the reference standard. The study adheres to STARD principles for diagnostic-accuracy research and uses predefined operating procedures for test execution, data capture, and analysis.

Study setting and workflow Participants are evaluated in the neuromuscular clinic of a tertiary hospital. The study uses a baseline-only design: all index and comparator tests are completed on the same day whenever feasible. A separate reliability session for image scoring occurs 48 hours to 7 days later without additional patient visits. The overall workflow is: (1) confirm eligibility and obtain consent; (2) complete standardized neurological examination and clinical scales; (3) perform or verify QST and SSR (irrespective of results); (4) perform WIWT; (5) acquire standardized fingertip photographs; (6) independent scoring of images by trained raters; (7) data entry and validation; (8) statistical analysis according to the prespecified plan.

Reference standard (composite) The reference standard integrates the treating neuromuscular specialist's judgment (history and examination) with at least one abnormal clinical scale among UENS or mTCNS using their published scoring rules. The scales are administered per their manuals by personnel trained on test instructions and scoring conventions. The reference standard classification (SFN vs no SFN) is recorded in a dedicated adjudication form. Test operators for WIWT, QST, and SSR do not have access to the reference classification at the time of testing.

Index test: WIWT-technical conduct Participants are seated upright. Both hands are immersed, at least to the distal interphalangeal crease, in water for 15 minutes. Before immersion, the skin is verified to be clean and completely dry. Hands are kept relaxed (neutral finger posture) and fingertips must not press against container surfaces. Because a thermostatically controlled bath is not available, immersion begins at 43-44 °C with expected passive cooling of approximately 2 °C every 5 minutes, targeting an end temperature of about 37-38 °C. Water temperature is measured with the service thermometer at 0, 5, 10 and 15 minutes to confirm the intended range. No water is added or replaced during immersion. A calibrated stopwatch is used to time the procedure. At completion, hands are gently patted dry and standardized photographs are obtained of the palmar distal phalanges of digits 2-5 of both hands. Environmental conditions are kept stable (indoor room, typical ambient temperature, indirect lighting) and recorded on the source form.

Image acquisition and standardization Photographs are taken with the clinic's digital camera or smartphone following a fixed template: (a) distance approximately 20-25 cm from fingertips; (b) camera aligned perpendicular to the palmar surface to minimize parallax; (c) neutral, diffuse illumination avoiding hard shadows; (d) inclusion of a 1-cm scale marker within the frame; (e) focus lock on the distal pad of each fingertip. Raw images are immediately reviewed for motion blur or framing errors and repeated if necessary before the participant leaves. Images are stored as high-resolution JPEG or HEIC (≥8 MP), transferred to the secure institutional drive, and automatically renamed by a deterministic convention (StudyID_Hand_Side_Digit_Timepoint.ext). No patient identifiers appear in filenames or image content.

Scoring rubric and rater training Wrinkling is graded on a 0-4 ordinal scale for digits 2-5 of each hand by trained raters who are not involved in the clinical reference assessment and are mutually blinded to QST/SSR results. Raters complete a short training using a curated set of example photographs with consensus labels, followed by a calibration exercise (≥20 images) with feedback until predefined agreement thresholds are met. For each participant, per-hand sums are computed and a bilateral summed score is derived; the bilateral classification threshold uses the prespecified rule (abnormal < 24; normal ≥ 24). For the reliability substudy, four raters independently score all images twice, separated by 48 hours to 7 days, with the second session presented in a randomized order to reduce recall. The image set used for the second session is identical to the first and contains no new photographs.

Comparator tests (QST and SSR) QST includes thermal detection thresholds and vibration thresholds measured with the clinic's standard equipment following manufacturer instructions and local laboratory SOPs, with device daily checks documented in the logbook. SSR is recorded from palmar electrodes with standard filter settings and sweep parameters; amplitude and latency are extracted according to laboratory conventions. Operators of QST and SSR are independent from the WIWT team and do not access the WIWT photographs or scores.

Bias mitigation and blinding To limit review and incorporation biases, the reference standard is defined a priori and does not include WIWT, QST, or SSR results. The WIWT examiner is masked to the reference classification and to QST/SSR readings; QST and SSR operators are masked to each other and to WIWT; image raters receive only coded image sets stripped of metadata. The order of WIWT versus QST/SSR is not fixed and is recorded to explore potential order effects. All analysis code and decision rules (for exclusions, tie handling, and outlier management) are prespecified.

Data collection and management Data are captured on paper case-report forms (CRFs) and transcribed into a REDCap-like electronic database hosted on the institutional server with user authentication, role-based access, and full audit trails. Double-data entry is applied to primary variables (reference classification, WIWT summed score, UENS/mTCNS totals); discrepancies are resolved by a third reviewer using the source documents. Automated data-validation rules check ranges (for example, temperature values at 0/5/10/15 minutes, test duration = 15 ± 1 min, score ranges 0-4 per digit), internal consistency (for example, bilateral sum equals the sum of component digits), and logical constraints (for example, no missing both "start temperature" and "end temperature"). A data dictionary defines variable names, formats, allowable codes, derivations, and edit checks. Versioning is handled at the database level; all changes after database lock require change-control approval and generate an audit entry.

Sample size rationale The planned sample size is approximately 30 participants, selected to provide acceptable precision for sensitivity and specificity estimates under plausible operating characteristics (for example, sensitivity ~0.80 and specificity ~0.70) with two-sided 95% confidence intervals of roughly ±0.10 under anticipated case-mix. The final sample size also accommodates the reliability substudy, ensuring that the number of images and raters provides adequate precision for intraclass correlation coefficients (ICCs) with confidence-interval widths ≤0.15 under expected variance components.

Statistical analysis overview Analyses are prespecified. For the primary diagnostic-accuracy analysis, WIWT is evaluated against the composite reference standard. Sensitivity, specificity, and their exact or 95% confidence intervals are reported at the prespecified bilateral sum threshold. ROC analysis treats the bilateral summed WIWT score as a continuous predictor; AUC and 95% CI are computed using non-parametric methods. Positive and negative predictive values are reported at the observed prevalence. Inter-rater reliability for the bilateral summed score uses a two-way random-effects, absolute-agreement ICC [ICC(2,1)], and intra-rater reliability uses a two-way mixed-effects ICC [ICC(3,1)] with 95% confidence intervals derived from ANOVA variance components; secondary reliability metrics (weighted kappa for ordinal per-digit grades) may be reported descriptively. Prespecified sensitivity analyses include: (a) exclusion of protocol-deviant WIWT runs (temperature/time deviations); (b) alternative temperature-window definitions; and (c) alternative classification cut-points explored descriptively without redefining the primary analysis. No hypothesis testing for between-test differences is required for the primary objective; if performed, comparisons of AUCs will use DeLong's method.

Data governance, confidentiality, and archiving All study data are de-identified at the point of storage; linkage files mapping StudyID to personal identifiers reside in a separate restricted directory accessible only to the clinical team. Photographs do not contain faces or unique marks beyond fingertip skin; rings and nail polish are removed when possible. Data are retained for the period required by institutional policy and local regulations. Access to the final analytic dataset and code is restricted to the analysis team; requests for de-identified data after publication follow the data-sharing statement entered elsewhere in the record.

Risk assessment and safety reporting WIWT, QST, and SSR are non-invasive procedures with minimal risk (primarily transient discomfort or skin maceration). Adverse events related to testing are expected to be rare and mild; any unexpected events temporally related to test execution are documented in the source forms and reported per institutional policy. The study does not use a formal data monitoring committee given its minimal-risk, non-interventional design.

Study timeline Recruitment is ongoing. Baseline testing and image acquisition occur on the day of enrollment; reliability scoring occurs within 48 hours to 7 days. Database lock is planned shortly after the anticipated primary completion date. The record will be updated as major milestones are reached (for example, changes in enrollment target, completion dates, or analysis plan).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Suspicion of small-fiber neuropathy based on history and/or physical examination by a neuromuscular neurology specialist.
* Sensory and motor nerve conduction studies within normal limits.
* Prior QST performed, regardless of result.
* Prior SSR performed, regardless of result.

Exclusion Criteria:

* Patients under 18 years.
* Individuals who do not wish to participate in the study or who decline informed consent.
* Patients with any contraindication to any of the aforementioned studies.
* Neurophysiological studies demonstrating large-fiber involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults evaluated at the Neuromuscular Department and Neurophysiology Laboratory of Hospital Británico de Buenos Aires (Argentina), a tertiary referral center. The source population includes consecutive clinic patients referred for assessment of suspected small-fiber neuropathy and healthy adult volunteers recruited from the hospital community. Recruitment occurs during routine outpatient activity; all index/comparator testing is performed on site.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of WIWT (%) vs composite reference (clinical + UENS/mTCNS abnormality) | Baseline (single visit; same-day completion of all tests)
  WIWT scoring: Each fingertip (digits 2-5 of both hands) is graded 0-4 after immersion (0 = no wrinkling; 4 = marked wrinkling). Per-hand sum 0-16; bilateral sum 0-32 (higher = more wrinkling/normal sympathetic function). Threshold to define test result: bilateral sum <24 = abnormal, ≥24 = normal.
  Procedure: Hands immersed 15 min, starting 43-44 °C with passive cooling ≈2 °C/5 min to ~37-38 °C; temperature checked at 0, 5, 10 min; no water added or replaced; standardized photographs scored by blinded raters.
  Reference standard: Neuromuscular specialist clinical assessment plus abnormality on ≥1 validated scale (UENS or mTCNS).
  Metrics: Sensitivity = TP/(TP+FN); Specificity = TN/(TN+FP); both reported as percent (%) with 95% CIs.

SECONDARY OUTCOMES:
ROC Area Under the Curve (AUC) for WIWT | Baseline
  ROC curve of WIWT (continuous summed score) vs. reference standard; AUC with 95% CI using non-parametric methods.
Positive and Negative Predictive Values (PPV, NPV) of WIWT | Baseline
  PPV = TP/(TP+FP); NPV = TN/(TN+FN) with 95% CIs at observed SFN prevalence in the study sample.
Inter-rater Reliability of WIWT Wrinkle Scoring (ICC) | Within 7 days (two image-rating sessions separated by 48 h-7 days).
  Four trained raters score standardized fingertip photographs; ICC(2,1), absolute agreement for summed wrinkle scores (digits 2-5 per hand; bilateral sum).
Intra-rater Reliability of WIWT Wrinkle Scoring (ICC) | 48 h-7 days between sessions.
  Same rater re-scores identical image set; ICC(3,1)
Comparative Diagnostic Performance: WIWT vs QST and SSR (AUC, Se/Sp) | Baseline
  At baseline, for each test (WIWT, QST, SSR) ROC curves are constructed against the composite reference (specialist assessment + abnormal UENS or mTCNS). AUCs with 95% CIs are reported and pairwise AUC comparisons (WIWT vs QST; WIWT vs SSR; QST vs SSR). Using prespecified thresholds-WIWT bilateral sum <24 = abnormal; QST abnormal per laboratory normative cut-offs; SSR abnormal if absent -we compute sensitivity and specificity (%, 95% CIs).

CONTACTS AND LOCATIONS:
Overall Officials: Lucas A Piedrafita Vico, MD, Principal Investigator — Hospital Británico de Buenos Aires
Locations (1):
- Hospital Britanico de Buenos Aires, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual data underlying the primary results may be shared upon reasonable request after publication for 36 months; data dictionary and analytic code available on request.

REFERENCES:
- [Background] Piedrafita Vico LA, Reisin R, Gonorazky S. Teaching NeuroImage: Absence of Wrinkles in Small Fiber Neuropathy. Neurology. 2022 Nov 22;99(21):962-963. doi: 10.1212/WNL.0000000000201320. Epub 2022 Sep 13. No abstract available. PMID 36100436
- [Background] Clark CV, Pentland B, Ewing DJ, Clarke BF. Decreased skin wrinkling in diabetes mellitus. Diabetes Care. 1984 May-Jun;7(3):224-7. doi: 10.2337/diacare.7.3.224. PMID 6734390
- [Background] Braham J, Sadeh M, Sarova-Pinhas I. Skin wrinkling on immersion of hands: a test of sympathetic function. Arch Neurol. 1979 Feb;36(2):113-4. doi: 10.1001/archneur.1979.00500380083013. PMID 420620
- [Background] Teoh HL, Chow A, Wilder-Smith EP. Skin wrinkling for diagnosing small fibre neuropathy: comparison with epidermal nerve density and sympathetic skin response. J Neurol Neurosurg Psychiatry. 2008 Jul;79(7):835-7. doi: 10.1136/jnnp.2007.140947. Epub 2008 Feb 12. PMID 18270233
- [Background] Wilder-Smith EP, Guo Y, Chow A. Stimulated skin wrinkling for predicting intraepidermal nerve fibre density. Clin Neurophysiol. 2009 May;120(5):953-8. doi: 10.1016/j.clinph.2009.03.011. Epub 2009 Apr 16. PMID 19375384
- [Background] Wilder-Smith EP. Stimulated skin wrinkling as an indicator of limb sympathetic function. Clin Neurophysiol. 2015 Jan;126(1):10-6. doi: 10.1016/j.clinph.2014.08.007. Epub 2014 Sep 2. PMID 25216595
- [Background] Cales L, Weber RA. Effect of water temperature on skin wrinkling. J Hand Surg Am. 1997 Jul;22(4):747-9. doi: 10.1016/s0363-5023(97)80141-4. PMID 9260639
- [Background] Singleton JR, Bixby B, Russell JW, Feldman EL, Peltier A, Goldstein J, Howard J, Smith AG. The Utah Early Neuropathy Scale: a sensitive clinical scale for early sensory predominant neuropathy. J Peripher Nerv Syst. 2008 Sep;13(3):218-27. doi: 10.1111/j.1529-8027.2008.00180.x. PMID 18844788
- [Background] Abraham A, Barnett C, Katzberg HD, Lovblom LE, Perkins BA, Bril V. Toronto Clinical Neuropathy Score is valid for a wide spectrum of polyneuropathies. Eur J Neurol. 2018 Mar;25(3):484-490. doi: 10.1111/ene.13533. Epub 2017 Dec 26. PMID 29194856
- [Background] Galosi E, Falco P, Di Pietro G, Leone C, Esposito N, De Stefano G, Di Stefano G, Truini A. The diagnostic accuracy of the small fiber neuropathy symptoms inventory questionnaire (SFN-SIQ) for identifying pure small fiber neuropathy. J Peripher Nerv Syst. 2022 Dec;27(4):283-290. doi: 10.1111/jns.12513. Epub 2022 Oct 5. PMID 36175394
- [Background] Bril V, Tomioka S, Buchanan RA, Perkins BA; mTCNS Study Group. Reliability and validity of the modified Toronto Clinical Neuropathy Score in diabetic sensorimotor polyneuropathy. Diabet Med. 2009 Mar;26(3):240-6. doi: 10.1111/j.1464-5491.2009.02667.x. PMID 19317818
- [Background] Zilliox LA, Ruby SK, Singh S, Zhan M, Russell JW. Clinical neuropathy scales in neuropathy associated with impaired glucose tolerance. J Diabetes Complications. 2015 Apr;29(3):372-7. doi: 10.1016/j.jdiacomp.2015.01.011. Epub 2015 Feb 3. PMID 25690405
- [Background] Novak P. Electrochemical skin conductance: a systematic review. Clin Auton Res. 2019 Feb;29(1):17-29. doi: 10.1007/s10286-017-0467-x. Epub 2017 Sep 26. PMID 28951985
- [Background] Terkelsen AJ, Karlsson P, Lauria G, Freeman R, Finnerup NB, Jensen TS. The diagnostic challenge of small fibre neuropathy: clinical presentations, evaluations, and causes. Lancet Neurol. 2017 Nov;16(11):934-944. doi: 10.1016/S1474-4422(17)30329-0. PMID 29029847
- [Background] Devigili G, Rinaldo S, Lombardi R, Cazzato D, Marchi M, Salvi E, Eleopra R, Lauria G. Diagnostic criteria for small fibre neuropathy in clinical practice and research. Brain. 2019 Dec 1;142(12):3728-3736. doi: 10.1093/brain/awz333. PMID 31665231
- [Background] Gendre T, Lefaucheur JP, Nordine T, Baba-Amer Y, Authier FJ, Devaux J, Creange A. Characterizing Acute-Onset Small Fiber Neuropathy. Neurol Neuroimmunol Neuroinflamm. 2024 Mar;11(2):e200195. doi: 10.1212/NXI.0000000000200195. Epub 2024 Jan 3. PMID 38170952
- [Background] Devigili G, Cazzato D, Lauria G. Clinical diagnosis and management of small fiber neuropathy: an update on best practice. Expert Rev Neurother. 2020 Sep;20(9):967-980. doi: 10.1080/14737175.2020.1794825. Epub 2020 Jul 23. PMID 32654574

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT07255573/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT07255573/ICF_001.pdf